CLINICAL TRIAL: NCT06975371
Title: Real-World Outcomes of Patients With HR-Positive HER2-Negative Metastatic Breast Cancer After Treatment With First-Line ET+CDK4/6i in the United States
Brief Title: Real-World Outcomes of Patients With Metastatic Breast Cancer After Treatment With First-Line ET+CDK4/6i
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: U31402-0012-NIS-MA
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Advanced/Metastatic HER2-negative Breast Cancer
Keywords: HR-positive; HER2-negative; Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HR+/HER2- metastatic breast cancer: Adults in the Flatiron database who are diagnosed with HR+/HER2- metastatic breast cancer and initiated a subsequent line of therapy (i.e., 2L) after progressing on 1L treatment with ET+CDK4/6i.
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — No study drug was administered in this non-interventional study.

SUMMARY:
This study aims to assess the treatment patterns and real-world outcomes of HR+/HER- metastatic breast cancer patients who have progressed on 1L ET + CDK4/6i and started a second line (2L) treatment within a real-world cohort in the United States Flatiron Health Database.

DETAILED DESCRIPTION:
This analysis will assess real-world outcomes in HR+/HER2- mBC patients who initiated a subsequent line of therapy (LOT) (i.e., 2L) after progressing on 1L treatment with ET+CDK4/6i. This study will also characterize the treatment patterns, clinical characteristics, and outcomes in this patient population. No study drug was administered in this non-interventional study.

ELIGIBILITY:
Inclusion criteria

* Patients with evidence of Stage IV or recurrent mBC with a metastatic diagnosis date on or after January 1, 2017
* Aged ≥18 years at mBC diagnosis date
* Received 1L ET + CDK 4/6i, with no other systemic agents, in the metastatic setting
* Had evidence of a rwP event during 1L ET + CDK 4/6i
* Evidence of a subsequent LOT following 1L ET + CDK 4/6i (start date of subsequent LOT = index treatment date)
* A record of HR+ status in the closest estrogen receptor (ER) or progesterone receptor (PR) test result occurring prior to or within 30 days after the index treatment date
* A record of HER2- status in the closest HER2 test result recorded prior to or on the index treatment date
* Index treatment date occurring at least 90 days prior to end of study period (30Sep2024)

Exclusion Criteria

• A record of estrogen receptor 1 (ESR1), phosphatidylinositol4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA), V-akt murine thymoma viral oncogene homolog (AKT1), phosphatase and tensin homolog (PTEN), or germline breast cancer gene (gBRCA) alteration/mutation prior to or within 30 days after index treatment date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort consists of adults in the Flatiron database who are diagnosed with HR+/HER2- mBC and initiated a subsequent LOT (i.e., 2L) after progressing on 1L treatment with ET+CDK4/6i.
Sampling Method: Non-Probability Sample
Enrollment: 1415 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Real-world progression-free survival (rwPFS) | Baseline up to end of observation period, approximately 7 years 9 months
  Real-world progression-free survival (rwPFS) will be calculated as the time from the index treatment date to the date of the first documented rwP event occurring >14 days after the index treatment date or date of death, whichever occurs first.

SECONDARY OUTCOMES:
Real-world overall survival (rwOS) | Baseline up to end of observation period, approximately 7 years 9 months
  Real-world overall survival (rwOS) will be calculated as the time from the index treatment date to death. Patients who do not experience the event of interest (death) will be censored at their last confirmed activity date.
Real-world time to discontinuation or death (rwTTD/D) | Baseline up to end of observation period, approximately 7 years 9 months
  Real-world time to treatment discontinuation or death (rwTTD/D) will be calculated for the index LOT. For the set of drugs contained in the index LOT, rwTTD/D will be calculated as the time from the first drug episode to the last drug episode or death, whichever comes first.
Real-world time to next treatment or death (rwTTNT/D) | Baseline up to end of observation period, approximately 7 years 9 months
  Real-world time to next treatment or death (rwTTNT/D) will be calculated for the index LOT as the time from the start of the LOT to the initiation of next LOT or death, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Director, Study Director — Daiichi Sankyo
Locations (1):
- Flatiron Health, Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No